CLINICAL TRIAL: NCT07043855
Title: Duration of Perioperative Antibiotic Prophylaxis in Patients Undergoing Pancreatoduodenectomy: a Randomized Controlled Trial
Brief Title: Duration of Perioperative Antibiotics in Pancreatoduodenectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-0529
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Pancreatoduodenectomy; PPPD; Infectious Complications
Keywords: preoperative antibiotics; perioperative antibiotics; prophylactic antibiotics
MeSH Terms: interventions — Cefazolin; Cefotaxime; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- single dose preoperative antibiotic (Experimental): Single Preoperative Dose of Cefazolin
  Interventions: Drug: single dose preoperative antibiotic
- prolonged perioperative antibiotics (Active Comparator): Preoperative Single-Dose Cefoxitin followed by Three-Day Cefotaxime and Metronidazole Prophylaxis
  Interventions: Drug: Prolonged perioperative antibiotics

INTERVENTIONS:
Drug: single dose preoperative antibiotic — Arm A is a single preoperative dose of cefazolin administered immediately before surgery
  Other Names: cefazolin
  Arms: single dose preoperative antibiotic
Drug: Prolonged perioperative antibiotics — Preoperative Single-Dose Cefoxitin followed by Three-Day Cefotaxime and Metronidazole Prophylaxis
  Other Names: cefoxitin followed by 3-day cefotaxime plus metronidazole
  Arms: prolonged perioperative antibiotics

SUMMARY:
The goal of this clinical trial is to learn if different prophylactic antibiotic regimens can prevent surgical site infections in adult patients undergoing pancreatoduodenectomy. The main questions it aims to answer are:

Does a single preoperative dose of cefazolin reduce the risk of surgical site infection? Does a three-day combination of cefotaxime plus metronidazole reduce the risk of surgical site infection? Researchers will compare a single dose of cefazolin to a three-day course of cefotaxime + metronidazole to see if there is a difference in postoperative infection rates.

Participants will:

* Be randomly assigned to one of two antibiotic regimens before and after surgery
* Receive either Arm A: one dose of cefazolin immediately before surgery Arm B: cefoxitin for perioperative antibiotics followed by cefotaxime plus metronidazole administered for three days after surgery
* Undergo routine postoperative monitoring for signs of infection
* Have any surgical site infections and related complications recorded until 30 days after surgery

DETAILED DESCRIPTION:
1. Brief background:

   Pancreaticoduodenectomy (PD) is one of the major hepatobiliopancreatic surgical procedures, with postoperative infectious complication rates reaching approximately 20-40%. International guidelines recommend a single preoperative dose of cefazolin as prophylactic antibiotic therapy for PD. However, due to concerns about high infectious complication rates, some institutions administer antibiotics for more than 24 hours postoperatively. This study aims to compare the surgical site infection rates between the internationally recommended single-dose cefazolin regimen and the current practice at Asan Medical Center of perioperative antibiotic prophylaxis consisting of preoperative second-generation cephalosporin (cefoxitin) administration followed by postoperative combined cefotaxime and metronidazole therapy for 3 days in patients undergoing PD. Through this comparison, we seek to contribute to establishing effective and safe antibiotic prophylaxis guidelines and advancing antimicrobial stewardship efforts for this patient population.

   //
2. Protocol summary:

This phase III, single-center randomized study at Seoul, Asan Medical Center will compare the efficacy of two antibiotic prophylaxis regimens in adult patients undergoing pancreatoduodenectomy. A total of 558 participants will be enrolled over a two-year period (from IRB approval), with follow-up through 30 days postoperatively. After informed consent and stratification by biliary stent status, patients will be randomized 1:1 to: (1) Intervention arm: single dose of cefazolin administered within 1 hour before skin incision. (2) Control (conventional) arm: Single dose of cefoxitin within 1 hour before skin incision, followed by cefotaxime plus metronidazole on postoperative days 1-3.

Participants will be assessed for surgical site infection (SSI) and other infectious complications. The primary outcome is the incidence of SSI within 30 days

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 18 to 80 years old scheduled for pancreaticoduodenectomy for any indication (including open, laparoscopic, and robotic surgery).
* Patients who have received sufficient explanation about this clinical trial and have voluntarily decided to participate and provided written informed consent.

Exclusion Criteria:

* History of Type 1 immediate hypersensitivity reaction to cefazolin, cefotaxime, or metronidazole.
* Active or uncontrolled infection prior to surgery for which treatment has not been completed.
* Use of antibiotics for any reason within 1 week prior to surgery.
* Long-term use of immunosuppressants due to other concomitant diseases.
* Undergoing dialysis or having renal dysfunction of KDIGO Grade 3 or higher (GFR < 45).
* Pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | within 30 days after PD/PPPD
  superficial/deep wound infection, organ-space infection

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD might not be shared

REFERENCES:
- [Background] Hwang DW, Kim HJ, Lee JH, Song KB, Kim MH, Lee SK, Choi KT, Jun IG, Bang JY, Kim SC. Effect of Enhanced Recovery After Surgery program on pancreaticoduodenectomy: a randomized controlled trial. J Hepatobiliary Pancreat Sci. 2019 Aug;26(8):360-369. doi: 10.1002/jhbp.641. Epub 2019 Jul 2. PMID 31152686
- [Background] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists (ASHP); Infectious Diseases Society of America (IDSA); Surgical Infection Society (SIS); Society for Healthcare Epidemiology of America (SHEA). Clinical practice guidelines for antimicrobial prophylaxis in surgery. Surg Infect (Larchmt). 2013 Feb;14(1):73-156. doi: 10.1089/sur.2013.9999. Epub 2013 Mar 5. No abstract available. PMID 23461695
- [Background] Boyev A, Arvide EM, Newhook TE, Prakash LR, Bruno ML, Dewhurst WL, Kim MP, Maxwell JE, Ikoma N, Snyder RA, Lee JE, Katz MHG, Tzeng CD. Prophylactic Antibiotic Duration and Infectious Complications in Pancreatoduodenectomy Patients With Biliary Stents: Opportunity for De-escalation. Ann Surg. 2024 Apr 1;279(4):657-664. doi: 10.1097/SLA.0000000000005982. Epub 2023 Jul 3. PMID 37389897
- [Background] D'Angelica MI, Ellis RJ, Liu JB, Brajcich BC, Gonen M, Thompson VM, Cohen ME, Seo SK, Zabor EC, Babicky ML, Bentrem DJ, Behrman SW, Bertens KA, Celinski SA, Chan CHF, Dillhoff M, Dixon MEB, Fernandez-Del Castillo C, Gholami S, House MG, Karanicolas PJ, Lavu H, Maithel SK, McAuliffe JC, Ott MJ, Reames BN, Sanford DE, Sarpel U, Scaife CL, Serrano PE, Smith T, Snyder RA, Talamonti MS, Weber SM, Yopp AC, Pitt HA, Ko CY. Piperacillin-Tazobactam Compared With Cefoxitin as Antimicrobial Prophylaxis for Pancreatoduodenectomy: A Randomized Clinical Trial. JAMA. 2023 May 9;329(18):1579-1588. doi: 10.1001/jama.2023.5728. PMID 37078771
- [Background] Sugawara G, Yokoyama Y, Ebata T, Mizuno T, Yagi T, Ando M, Nagino M. Duration of Antimicrobial Prophylaxis in Patients Undergoing Major Hepatectomy With Extrahepatic Bile Duct Resection: A Randomized Controlled Trial. Ann Surg. 2018 Jan;267(1):142-148. doi: 10.1097/SLA.0000000000002049. PMID 27759623
- [Background] Yamamoto T, Satoi S, Fujii T, Yamada S, Yanagimoto H, Yamaki S, Takami H, Hirooka S, Kosaka H, Kotsuka M, Miyara T, Kodera Y. Dual-center randomized clinical trial exploring the optimal duration of antimicrobial prophylaxis in patients undergoing pancreaticoduodenectomy following biliary drainage. Ann Gastroenterol Surg. 2018 Sep 17;2(6):442-450. doi: 10.1002/ags3.12209. eCollection 2018 Nov. PMID 30460348
- [Background] Okamura K, Tanaka K, Miura T, Nakanishi Y, Noji T, Nakamura T, Tsuchikawa T, Okamura K, Shichinohe T, Hirano S. Randomized controlled trial of perioperative antimicrobial therapy based on the results of preoperative bile cultures in patients undergoing biliary reconstruction. J Hepatobiliary Pancreat Sci. 2017 Jul;24(7):382-393. doi: 10.1002/jhbp.453. Epub 2017 May 6. PMID 28371248